CLINICAL TRIAL: NCT04711473
Title: Choice Architecture and Mailed Colorectal Cancer Screening Outreach in a Community Health Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Principal Investigator, Shivan Mehta, Principal Investigator, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UPCC 13220; 843772 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer
Keywords: screening; prevention; colonoscopy; stool testing
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Colonoscopy Only (Active Comparator): Participants in this arm will receive a letter from their provider informing them they are overdue for colon cancer screening and requesting their participation in colonoscopy, and including a referral for the procedure at a local endoscopy center. Participants will be provided a phone number if interested in navigated colonoscopy scheduling.
  Interventions: Behavioral: Colonoscopy Only
- Choice (Experimental): Participants in this arm will receive a letter from their provider informing them they are overdue for colon cancer screening and requesting their participation in their choice of either colonoscopy or mailed fecal immunochemical testing (FIT). The letter will include both a referral for the colonoscopy at a local endoscopy enter and a FIT kit with a lab requisition and instructions for completion.
  Interventions: Behavioral: Choice
- FIT Only (Experimental): Participants in this arm will receive a letter from their provider informing them they are overdue for colon cancer screening and requesting their participation in FIT testing. The letter will include a FIT kit with lab requisition and instructions for completion.
  Interventions: Behavioral: FIT Only

INTERVENTIONS:
Behavioral: Colonoscopy Only — Mailed letter asking participants to complete CRC screening by colonoscopy
  Arms: Colonoscopy Only
Behavioral: Choice — Mailed letter and FIT test asking participants to complete CRC screening by their choice of either colonoscopy or mailed FIT
  Arms: Choice
Behavioral: FIT Only — Mailed letter and FIT test asking participants to complete CRC screening by mailed FIT
  Arms: FIT Only

SUMMARY:
This is a 3-arm randomized trial aimed at increasing rates of participation in colorectal cancer (CRC) screening by outreach to patients' homes using choice architecture informed by behavioral science principles.

DETAILED DESCRIPTION:
The investigators will evaluate the effectiveness of mailed outreach with choice between colonoscopy and FIT, and FIT alone, as compared to colonoscopy alone in increasing CRC screening rates.

ELIGIBILITY:
Inclusion Criteria:

1. At least 1 visit with CHDC in the past 2 years
2. Not up to date on CRC screening (no evidence of colonoscopy in the last 10 years, sigmoidoscopy in the last 5 years, or stool testing in the past 12 months)

Exclusion Criteria:

1. History of CRC or polyps
2. Significant family history of CRC
3. History of Inflammatory Bowel Disease or Ulcerative Colitis
4. History of colectomy
5. History of metastatic cancer
6. Current use of Medication Assisted Therapy (MAT)

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Colorectal Cancer Screening Completion | 6 months from initial outreach
  Screening completion rate in arm 2 (Choice) to arm 1 (Colonoscopy only) and arm 3 (FIT only) separately.

SECONDARY OUTCOMES:
Choice of Colorectal Cancer Screening Test | 6 months from initial outreach
  The proportion of patients choosing either FIT or Colonoscopy in study arm 2 (Choice)

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Community Health and Dental Care, Pottstown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta SJ, Palat S, McDonald C, Reitz C, Okorie E, Williams K, Tao J, Shaw PA, Glanz K, Asch DA. A Randomized Trial of Choice Architecture and Mailed Colorectal Cancer Screening Outreach in a Community Health Setting. Clin Gastroenterol Hepatol. 2024 Oct;22(10):2117-2124.e2. doi: 10.1016/j.cgh.2024.04.003. Epub 2024 Apr 30. PMID 38697235